CLINICAL TRIAL: NCT00188656
Title: Minimum Dose CT in the Detection of Lung Nodules in Patients With Head and Neck Cancer
Brief Title: Computed Tomography (CT) in Head and Neck Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: insufficient recruitment
Sponsor: University Health Network, Toronto (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 03-0467
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2010-12-15 (Estimated); Status verified 2010-12

CONDITIONS: Lung Tumors
MeSH Terms: conditions — Lung Neoplasms

INTERVENTIONS:
Procedure: CT thorax

SUMMARY:
This study is conducting a comparison of chest x-ray (CXR) and minimum dose thoracic CT (MnDCT) in the detection of lung nodules (metastases) in patients with head and neck carcinoma.

DETAILED DESCRIPTION:
A comparison of chest x-ray (CXR) and minimum dose thoracic CT (MnDCT)in the detection of lung nodules (metastases) in patients with head and neck carcinoma

ELIGIBILITY:
Inclusion Criteria:

* Patients with squamous cell carcinoma of the head and neck

Exclusion Criteria:

* None

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2003-08; Study Completion 2006-09

PRIMARY OUTCOMES:
Detection of lung metastases

CONTACTS AND LOCATIONS:
Overall Officials: Narinder Paul, FRCP C, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada